CLINICAL TRIAL: NCT00168805
Title: RE-MODEL (Thromboembolism Prevention After Knee Surgery). Two Different Dose Regimens of Orally Administered Dabigatran Etexilate Capsules [150 or 220 mg Once Daily Starting With a Half Dose (i.e.75 or 110 mg) on the Day of Surgery] Compared to Subcutaneous Enoxaparin 40 mg Once Daily for 6-10 Days
Brief Title: RE-MODEL Dabigatran Etexilate 150mg or 220mg Once Daily (o.d.) Versus (v.s.) Enoxaparin 40mg o.d. for Prevention of Thrombosis After Knee Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.25; 2004-001317-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-02

CONDITIONS: Arthroplasty, Replacement, Knee; Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Enoxaparin; Dabigatran

ARMS (3):
- dabigatran etexilate 220 mg (Experimental): 220 mg once daily
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate 150 mg (Experimental): 150 mg once daily
  Interventions: Drug: dabigatran etexilate
- enoxaparin (Active Comparator): 40 mg once daily
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: enoxaparin — 40 mg once daily
  Arms: enoxaparin
Drug: dabigatran etexilate — 150 mg once daily
  Arms: dabigatran etexilate 150 mg
Drug: dabigatran etexilate — 220 mg once daily
  Arms: dabigatran etexilate 220 mg

SUMMARY:
A phase III, randomised, parallel-group, double-blind, active controlled study to investigate the ef ficacy and safety of two different dose regimens of orally administered dabigatran etexilate capsule s [150 or 220 mg once daily starting with a half dose (i.e.75 or 110 mg) on the day of surgery] comp ared to subcutaneous enoxaparin 40 mg once daily for 6 to 10 days, in prevention of venous thromboem bolism in patients with primary elective total knee replacement surgery. RE-MODEL (Thromboembolism prevention after knee surgery)

ELIGIBILITY:
Inclusion criteria

Inclusion criteria (selected):

* Patients (18 years or older) scheduled to undergo a primary, unilateral, elect ive total knee replacement
* Written Informed Consent

Exclusion criteria

Exclusion criteria (selected):

* Patients with an excessive risk of bleeding, for example because of history of bleeding diathesis major surgery or trauma within the last 3 months history of haemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm, arteriovenous (AV) malformation or aneurysm clinically relevant bleeding or gastric / duodenal ulcer within the last 6 months treatment with anticoagulants within 7 days prior to joint replacement surgery or anticipated need during the study treatment period thrombocytopenia.
* Active malignant disease or current cytostatic treatment
* Known severe renal insufficiency
* Liver disease expected to have any potential impact on survival, or elevated aspartate aminotransferase (AST) or alanine transaminase (ALT) > 2x upper limit of normal
* Recent unstable cardiovascular disease or history of myocardial infarction within the last 3 months
* Pre-menopausal women who are pregnant or nursing, or are of child-bearing pote ntial and are not practising or do not plan to continue practising acceptable me thods of birth control
* Allergy to radio opaque contrast media or iodine, heparins (incl. heparin indu ced thrombocytopenia) or dabigatran
* Contraindications to enoxaparin
* Participation in a clinical trial during the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2101 (Actual)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (105):
- Australia (12):
  - 1160.25.06108 Boehringer Ingelheim Investigational Site, Garren, Australian Capital Territory
  - 1160.25.06106 Boehringer Ingelheim Investigational Site, Kogarah, New South Wales
  - 1160.25.06110 Boehringer Ingelheim Investigational Site, Lismore, New South Wales
  - 1160.25.06105 Boehringer Ingelheim Investigational Site, Bedford Park, South Australia
  - 1160.25.06107 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 1160.25.06109 Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - 1160.25.06104 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.25.06102 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1160.25.06101 Boehringer Ingelheim Investigational Site, Malvern, Victoria
  - 1160.25.06103 Boehringer Ingelheim Investigational Site, Ringwood East, Victoria
  - 1160.25.06113 Boehringer Ingelheim Investigational Site, Windsor, Victoria
  - 1160.25.06111 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Austria (4):
  - 1160.25.04304 Boehringer Ingelheim Investigational Site, Linz
  - 1160.25.04302 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.25.04303 Boehringer Ingelheim Investigational Site, Wels
  - 1160.25.04301 Boehringer Ingelheim Investigational Site, Wiener Neustadt
- Belgium (8):
  - 1160.25.03207 UVC Brugmann, Brussels
  - 1160.25.03209 ZOL St. Jan, Genk
  - 1160.25.03206 Campus Sint-Lucas, Ghent
  - 1160.25.03208 UZ Gent, Ghent
  - 1160.25.03202 Virga Jesseziekenhuis, Hasselt
  - 1160.25.03203 AZ Sint Elisabeth, Herentals
  - 1160.25.03205 Ziekenhuis Oost-Limburg, Lanaken
  - 1160.25.03201 UZ Gasthuisberg, Leuven
- Czechia (9):
  - 1160.25.42004 Boehringer Ingelheim Investigational Site, Brno-Bohunice
  - 1160.25.42010 Boehringer Ingelheim Investigational Site, Chomutov
  - 1160.25.42009 Boehringer Ingelheim Investigational Site, Havlíčkův Brod
  - 1160.25.42002 Boehringer Ingelheim Investigational Site, Kladno
  - 1160.25.42006 Boehringer Ingelheim Investigational Site, Kolín
  - 1160.25.42003 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.25.42001 Boehringer Ingelheim Investigational Site, Pilsen
  - 1160.25.42007 Boehringer Ingelheim Investigational Site, Pradubice
  - 1160.25.42005 Boehringer Ingelheim Investigational Site, Prague
- Denmark (5):
  - 1160.25.04571 Boehringer Ingelheim Investigational Site, Hellerup
  - 1160.25.04570 Boehringer Ingelheim Investigational Site, Hørsholm
  - 1160.25.04573 Boehringer Ingelheim Investigational Site, København NV
  - 1160.25.04574 Boehringer Ingelheim Investigational Site, København S
  - 1160.25.04575 Boehringer Ingelheim Investigational Site, Silkeborg
- Finland (4):
  - 1160.25.35803 Boehringer Ingelheim Investigational Site, Helsinki
  - 1160.25.35802 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.25.35801 Boehringer Ingelheim Investigational Site, Oulu
  - 1160.25.35804 Boehringer Ingelheim Investigational Site, Seinäjoki
- France (9):
  - 1160.25.03304 Boehringer Ingelheim Investigational Site, Amiens
  - 1160.25.03307 Boehringer Ingelheim Investigational Site, Annecy
  - 1160.25.03305 Boehringer Ingelheim Investigational Site, La Rochelle
  - 1160.25.03301 Boehringer Ingelheim Investigational Site, Paris
  - 1160.25.03306 Boehringer Ingelheim Investigational Site, Poitiers
  - 1160.25.03303 Boehringer Ingelheim Investigational Site, Roubaix
  - 1160.25.03309 Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.25.03302 Boehringer Ingelheim Investigational Site, Soyaux
  - 1160.25.03308 Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (9):
  - 1160.25.04906 Caritaskrankenhaus, Bad Mergentheim
  - 1160.25.04910 F.-A.-Universität Erlangen-Nürnberg, Erlangen
  - 1160.25.04904 Orthopädische Universitätsklinik, Frankfurt
  - 1160.25.04902 Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - 1160.25.04911 Martin-Luther-Universität Halle-Wittenberg, Halle
  - 1160.25.04912 Orthopädische Klinik Markgröningen gGmbH, Markgröningen
  - 1160.25.04901 Kreiskrankenhaus, Rheinfelden
  - 1160.25.04903 Hellmuth-Ulrici-Kliniken, Sommerfeld
  - 1160.25.04905 Aukammklinik, Wiesbaden
- Hungary (6):
  - 1160.25.03607 Boehringer Ingelheim Investigational Site, Békéscsaba
  - 1160.25.03603 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.25.03601 Boehringer Ingelheim Investigational Site, Gyula
  - 1160.25.03604 Boehringer Ingelheim Investigational Site, Kecskemét
  - 1160.25.03602 Boehringer Ingelheim Investigational Site, Szeged
  - 1160.25.03605 Boehringer Ingelheim Investigational Site, Székesfehérvár
- Italy (6):
  - 1160.25.03906 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.25.03905 Boehringer Ingelheim Investigational Site, Parma
  - 1160.25.03901 Boehringer Ingelheim Investigational Site, Pavia
  - 1160.25.03903 Boehringer Ingelheim Investigational Site, Piacenza
  - 1160.25.03904 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1160.25.03902 Boehringer Ingelheim Investigational Site, Treviso
- Netherlands (6):
  - 1160.25.03102 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.25.03103 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.25.03101 Boehringer Ingelheim Investigational Site, Hoofddorp
  - 1160.25.03104 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1160.25.03105 Boehringer Ingelheim Investigational Site, Sittard
  - 1160.25.03106 Boehringer Ingelheim Investigational Site, Zwolle
- Poland (4):
  - 1160.25.04804 Boehringer Ingelheim Investigational Site, Kielce
  - 1160.25.04806 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.25.04807 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.25.04803 Boehringer Ingelheim Investigational Site, Warsaw
- South Africa (3):
  - 1160.25.02701 Boehringer Ingelheim Investigational Site, Bryanston
  - 1160.25.02703 Boehringer Ingelheim Investigational Site, Randburg
  - 1160.25.02702 Boehringer Ingelheim Investigational Site, Sandton
- Spain (11):
  - 1160.25.03405 Boehringer Ingelheim Investigational Site, Alcorcón (Madrid)
  - 1160.25.03403 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.25.03411 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.25.03407 Boehringer Ingelheim Investigational Site, Hospitalet (Barcelona)
  - 1160.25.03409 Boehringer Ingelheim Investigational Site, Jaén
  - 1160.25.03401 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.25.03402 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.25.03404 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.25.03406 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.25.03408 Boehringer Ingelheim Investigational Site, Móstoles (Madrid)
  - 1160.25.03410 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (9):
  - 1160.25.04602 Boehringer Ingelheim Investigational Site, Falköping
  - 1160.25.04601 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.25.04607 Boehringer Ingelheim Investigational Site, Halmstad
  - 1160.25.04603 Boehringer Ingelheim Investigational Site, Kungälv
  - 1160.25.04608 Boehringer Ingelheim Investigational Site, Lidköping
  - 1160.25.04605 Boehringer Ingelheim Investigational Site, Linköping
  - 1160.25.04604 Boehringer Ingelheim Investigational Site, Mölndal
  - 1160.25.04610 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.25.04609 Boehringer Ingelheim Investigational Site, Varberg

REFERENCES:
- [Derived] Eriksson BI, Dahl OE, Rosencher N, Clemens A, Hantel S, Kurth AA. Efficacy of delayed thromboprophylaxis with dabigatran: pooled analysis. Thromb Res. 2012 Dec;130(6):871-6. doi: 10.1016/j.thromres.2012.08.315. Epub 2012 Sep 17. PMID 22995531
- [Derived] Rosencher N, Noack H, Feuring M, Clemens A, Friedman RJ, Eriksson BI. Type of anaesthesia and the safety and efficacy of thromboprophylaxis with enoxaparin or dabigatran etexilate in major orthopaedic surgery: pooled analysis of three randomized controlled trials. Thromb J. 2012 Jun 18;10(1):9. doi: 10.1186/1477-9560-10-9. PMID 22709460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment period is from first administration of study medication, until 3 days after last administration of study medication. Treatment duration is planned for 8 days. The study period is from first administration of study medication until day 84 - 91.
Pre-assignment Details: Whilst 2101 patients were enrolled/randomised to treatment prior to surgery in this trial, only 2076 started treatment. Therefore, 25 patients were randomised but not treated (treatment was planned to start post surgery).
Groups:
- Dabigatran 220mg; Dabigatran 150mg: qd (once daily) oral
- Enoxaparin: 40mg qd (once daily) subcutaneous
Period: Overall Study
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 679 | 703 | 694
Completed | 608 | 625 | 616
Not Completed | 71 | 78 | 78
Not completed — Adverse Event | 7 | 11 | 16
Not completed — Protocol Violation | 12 | 11 | 8
Not completed — Lost to Follow-up | 12 | 17 | 11
Not completed — Withdrawal by Subject | 16 | 18 | 21
Not completed — Other | 24 | 21 | 22
Period: Treatment
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 679 | 703 | 694
Completed | 630 | 647 | 632
Not Completed | 49 | 56 | 62
Not completed — Adverse Event | 25 | 26 | 32
Not completed — Protocol Violation | 3 | 5 | 5
Not completed — Withdrawal by Subject | 3 | 7 | 8
Not completed — Other | 18 | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin | Total
Number analyzed (Participants) | 679 | 703 | 694 | 2076
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (9.0) | 67.5 (8.8) | 68.3 (8.8) | 67.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 441 | 451 | 478 | 1370
  Male | 238 | 252 | 216 | 706
Body Mass Index N=(677;702;692;2071) [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (4.9) | 30.1 (5.0) | 29.8 (4.9) | 29.9 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Venous Thromboembolic Event and All-cause Mortality During Treatment Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
  All of these components and all deaths were centrally adjudicated by the VTE events committee, which was not aware of the treatment allocation of the patients.
Time Frame: First administration until 6-10 days
Population: Full Analysis Set (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for distal and proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 503 | 526 | 512
Participants | 183 | 213 | 193
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — Non-inferiority Analysis with NI margin 9.2%. This results from the null-hypotheses of non-inferiority testing, where the absolute risk difference has to be below 9.2%. Non-inferiority can only be shown with CI; p = 0.6648, Normal approximation — p-value is for superiority testing; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.3, 95% CI [-7.3 to 4.6]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3553, Normal approximation — p-value is for superiority testing; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 2.8, 95% CI [-3.1 to 8.7]

2. Secondary Outcome: Number of Participants With Major Venous Thromboembolic Event and Venous Thromboembolic Event-related Mortality During Treatment Period
Description: Major Venous Thromboembolic Event (VTE) is defined as proximal DVT and PE, as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - major (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died by a Venous Thromboembolic Event-related death)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 506 | 527 | 511
Participants | 13 | 20 | 18
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.3760, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.0, 95% CI [-3.1 to 1.2]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.8151, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.3, 95% CI [-2.0 to 2.6]

3. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis During Treatment Period
Description: Proximal Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - pDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 506 | 525 | 510
Participants | 13 | 18 | 17
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.4715, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -0.8, 95% CI [-2.8 to 1.3]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.9325, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.1, 95% CI [-2.1 to 2.3]

4. Secondary Outcome: Number of Participants With Total Deep Vein Thrombosis During Treatment Period
Description: Total Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - tDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 503 | 524 | 511
Participants | 182 | 211 | 192
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.6463, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.4, 95% CI [-7.3 to 4.5]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.3740, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 2.7, 95% CI [-3.2 to 8.6]

5. Secondary Outcome: Number of Participants With Symptomatic Deep Vein Thrombosis During Treatment Period
Description: Symptomatic Deep Vein Thrombosis, confirmed by venous compression ultrasound, venography or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - op (all patients who are treated and operated)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 675 | 696 | 685
Participants | 1 | 3 | 8
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0385, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.1414, Fisher Exact

6. Secondary Outcome: Number of Participants With Pulmonary Embolism During Treatment Period
Description: Pulmonary embolism confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - op
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 675 | 696 | 685
Participants | 0 | 1 | 1
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact

7. Secondary Outcome: Number of Participants Who Died During Treatment Period
Description: All cause death, as adjudicated by the VTE events committee
Time Frame: First administration until 6-10 days
Population: Full Analysis Set - op
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 675 | 696 | 685
Participants | 1 | 1 | 1
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact

8. Secondary Outcome: Number of Participants With Total Venous Thromboembolic Event (VTE) and All-cause Mortality During the Follow-up Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
Time Frame: 3 months
Population: Patients with any data available during follow-up
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 658 | 679 | 665
Participants
  Total VTE and all-cause mortality | 4 | 3 | 2
  asymptotic Deep Vein Thrombosis | 0 | 1 | 0
  symptotic Deep Vein Thrombosis | 1 | 2 | 0
  Pulmonary Embolism | 2 | 0 | 0
  death | 1 | 0 | 2

9. Secondary Outcome: Number of Participants With Bleeding Events (Defined According to Modified McMaster Criteria) During Treatment Period
Description: Major bleeding events were defined as
  * fatal
  * clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected
  * clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected
  * symptomatic retroperitoneal, intracranial, intraocular or intraspinal
  * requiring treatment cessation
  * leading to re-operation
  Clinically-relevant was defined as
  * spontaneous skin hematoma greater than or equal to 25 cm²
  * wound hematoma greater than or equal to 100 cm²
  * spontaneous nose bleed lasting longer than 5 min
  * macroscopic hematuria spontaneous or lasting longer than 24 hours if associated with an intervention
  * spontaneous rectal bleeding (more than a spot on toilet paper)
  * gingival bleeding lasting longer than 5 min
  * any other bleeding event considered clinically relevant by the investigator
  Minor bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: First administration until 6-10 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 679 | 703 | 694
Participants
  Major | 10 | 9 | 9
  Clinically relevant | 40 | 48 | 37
  Minor | 60 | 59 | 69
  None | 569 | 587 | 579
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.8209, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 1.0000, Fisher Exact

10. Secondary Outcome: Blood Transfusion
Description: Blood transfusion for treated and operated patients on Day of surgery.
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 675 | 696 | 685
participants
  Patients with >=1 transfusions | 242 | 253 | 265
  Patients with >=1 non-autologous transfusions | 87 | 86 | 120

11. Secondary Outcome: Volume of Blood Loss
Description: Volume of blood loss for treated and operated patients during surgery.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 650 | 669 | 658
mL | 187 (258) | 190 (250) | 191 (254)

12. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: First administration to end of study
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 621 | 645 | 637
participants
  AST increase N=(620;645;636) | 9 | 6 | 9
  AST decrease N=(620;645;636) | 0 | 0 | 0
  ALT increase N=(621;645;637) | 16 | 21 | 24
  ALT decrease N=(621;645;637) | 0 | 0 | 0
  Bilirubin increase N=(619;644;635) | 19 | 23 | 14
  Bilirubin decrease N=(619;644;635) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration to end of study
Description: Treatment emergent events (last medication + 3 days)
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 31/679 | 44/703 | 43/694
Other Adverse Events (participants affected / at risk) | 405/679 | 438/703 | 426/694
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=679) | Dabigatran 150mg (N=703) | Enoxaparin (N=694)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0
Drug ineffective (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0
Secretion discharge (General disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Postoperative infection (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 2 | 1
Body temperature increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Immobilisation prolonged (Social circumstances) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 13 | 9
Haematoma (Vascular disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 2
Wound haemorrhage (Vascular disorders) | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=679) | Dabigatran 150mg (N=703) | Enoxaparin (N=694)
Constipation (Gastrointestinal disorders) | 71 | 65 | 77
Diarrhoea (Gastrointestinal disorders) | 27 | 41 | 24
Nausea (Gastrointestinal disorders) | 136 | 138 | 173
Vomiting (Gastrointestinal disorders) | 112 | 113 | 118
Oedema peripheral (General disorders) | 50 | 55 | 52
Pyrexia (General disorders) | 54 | 64 | 62
Post procedural haematoma (Injury, poisoning and procedural complications) | 28 | 31 | 36
Insomnia (Psychiatric disorders) | 66 | 65 | 69
Deep vein thrombosis (Vascular disorders) | 78 | 106 | 89
Hypotension (Vascular disorders) | 19 | 37 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract